CLINICAL TRIAL: NCT00088140
Title: A Dose Response Study of a Caspase Inhibitor in Hepatitis C Patients
Brief Title: A Caspase Inhibitor in Chronic Hepatitis C (HCV) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Collaborators: Idun Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-000006556-PRO-0007
Record Dates: First submitted 2004-07-20; First posted 2004-07-21 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- IDN-6556 5 mg twice a day (BID) (Active Comparator)
  Interventions: Drug: IDN-6556
- IDN-6556 25mg twice a day (BID) (Active Comparator)
  Interventions: Drug: IDN-6556
- IDN-6556 50 mg twice a day (BID) (Active Comparator)
  Interventions: Drug: IDN-6556

INTERVENTIONS:
Drug: IDN-6556
  Arms: IDN-6556 25mg twice a day (BID); IDN-6556 5 mg twice a day (BID); IDN-6556 50 mg twice a day (BID)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if IDN-6556, when given orally, is safe and effective in patients with chronic hepatitis C virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection
* Unsuccessful prior HCV treatment
* Liver impairment (either AST or ALT 1.5-10.0 x ULN)
* Alpha-fetoprotein <= 50 ng/mL
* Adequate hematologic parameters

Exclusion Criteria:

* Decompensated or severe liver disease
* Hepatocellular carcinoma
* HIV infection
* Co-infection with hepatitis B virus (HBV)
* Renal impairment
* Pancreatitis
* Use of illicit or drugs of abuse
* History of alcohol abuse
* Presence of clinically significant cardiac arrhythmias
* If female, pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2004-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Median absolute change in aspartate transaminase (AST) values measured from baseline to Week 10
Median absolute change in alanine aminotransferase (ALT) values measured from baseline to Week 10

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scripps Clinic, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - The Mayo Clinic, Rochester, Minnesota
  - Mt. Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Medical College of Virginia, Richmond, Virginia